CLINICAL TRIAL: NCT01331096
Title: Tele-Anesthesia - Trans-Continental Anesthesia Compared to Standard Practice
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: Teleanesthesia3054
Record Dates: First submitted 2011-04-06; First posted 2011-04-07 (Estimated); Last update posted 2011-04-07 (Estimated); Status verified 2011-03

CONDITIONS: Thyroid Gland Resection
Keywords: thyroid gland resection surgery; total intravenous anesthesia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Anesthetic drugs manually administrated
- Automated anesthesia delivery system

SUMMARY:
Patients in Pisa will undergo thyroid gland surgery. In the protocol group anesthesia will be performed using an automated anesthesia delivery system; preoperative and intra-operative assessment of patients will be performed via video-conferencing from Montreal, which will also monitor and control anesthesia delivery via distant Internet connection - as supervision of functioning of the automated anesthesia delivery system. In the control group anesthesia will be performed in a standard fashion with manual control of the syringe pumps infusing anesthetics drugs.

The hypothesis is that Tele-anesthesia, considered as preoperative assessment and anesthetic control of an automated anesthesia delivery system is feasible and reliable via standard means of internet communication (distant control via virtual network) and performed as well or even better than manual control of the anesthetic drugs infusion.

ELIGIBILITY:
Inclusion Criteria:

* Elective patients
* Patient scheduled for surgery under spinal anesthesia
* Patients aged 18 to 85 years

Exclusion Criteria:

* Unable to provide informed consent
* Comatose patients
* Patients with dementia
* Allergy to Propofol

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective thyroid gland surgery
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-03

PRIMARY OUTCOMES:
Performance of closed-loop system for propofol administration, controlled remotely, compared with the performance of propofol manually administered to maintain in both case the level of hypnosis close to the BIS target. | 2 years
  Hypnosis is monitored during the surgery according to the brain activity values provided by an objective monitoring parameter, called Bispectral Index (BIS). A BIS target of 45 is aimed trough the surgery. Performance of propofol hypnosis will be determined clinically by recording the % of sedation time during which the actual BIS is within 10% of the target BIS (excellent control), within 11 -20% (good control), between 21-30% (fair control) and beyond 30% of target (inadequate control).

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy

REFERENCES:
- [Derived] Hemmerling TM, Arbeid E, Wehbe M, Cyr S, Giunta F, Zaouter C. Transcontinental anaesthesia: a pilot study. Br J Anaesth. 2013 May;110(5):758-63. doi: 10.1093/bja/aes498. Epub 2013 Mar 10. PMID 23479676